CLINICAL TRIAL: NCT00198835
Title: Evaluation Research of the Nutrition Interventions in the INHP II Areas of CARE India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H.22.03.06.02.A2
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2005-07

CONDITIONS: Underweight; Stunting; Wasting; Anemia
Keywords: malnutrition; anemia; infants; children; India
MeSH Terms: conditions — Thinness; Growth Disorders; Cachexia; Anemia; Malnutrition | interventions — Maternal Nutritional Physiological Phenomena

INTERVENTIONS:
Behavioral: Maternal nutrition and infant feeding advice

SUMMARY:
This study is designed to evaluate the effectiveness of CARE India's Integrated Nutrition and Health Program (INHP II) to reduce malnutrition among children 0-23 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with a child 0-23 months of age
* Children 0-23 months of age
* Currently pregnant women
* Resides in the program or control area

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17000
Dates: Start 2003-08 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of underweight among children 0-23 months
Prevalence of stunting among children 0-23 months
Prevalence of wasting among children 0-23 months
Prevalence of anemia among children 12-23 months

CONTACTS AND LOCATIONS:
Overall Officials: Michele L Dreyfuss, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- King George Medical University, Lucknow, Uttar Pradesh, India

REFERENCES:
- [Derived] Singh V, Ahmed S, Dreyfuss ML, Kiran U, Chaudhery DN, Srivastava VK, Ahuja RC, Baqui AH, Darmstadt GL, Santosham M, West KP Jr. An integrated nutrition and health program package on IYCN improves breastfeeding but not complementary feeding and nutritional status in rural northern India: A quasi-experimental randomized longitudinal study. PLoS One. 2017 Sep 20;12(9):e0185030. doi: 10.1371/journal.pone.0185030. eCollection 2017. PMID 28931088
- [Derived] Singh V, Ahmed S, Dreyfuss ML, Kiran U, Chaudhery DN, Srivastava VK, Ahuja RC, Baqui AH, Darmstadt GL, Santosham M, West KP Jr. Non-governmental organization facilitation of a community-based nutrition and health program: Effect on program exposure and associated infant feeding practices in rural India. PLoS One. 2017 Sep 14;12(9):e0183316. doi: 10.1371/journal.pone.0183316. eCollection 2017. PMID 28910328